CLINICAL TRIAL: NCT01385085
Title: Impact of Work Environment Absent of Natural Light on Vitamin D Levels
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Head of Industrial Hygiene, Occupational Medicine and Medical Classification Branch , IDF
Other Study IDs: 922-2010-IDF-CTIL
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Sunlight; Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No natural sunlight: one group works in a basement with no natural sunlight
- Low level of Natural Sunlight: the second group work in offices with unopenable windows.
- High level of Natural Sunlight: The third group works outdoors.

SUMMARY:
Three types of workers exposed to different levels of natural sunlight will be tested for Vitamin D blood level, PTH, Ca, P, albumin and alkaline phosphatase.

In addition, each tested worker will be asked to fill a questionnaire for demographic, medical and personal habit information.

ELIGIBILITY:
Inclusion Criteria:

* people employed in their current work place at least 6 months,

Exclusion Criteria:

* people who consume food additives containing Vitamin D.
* people who have a chronic illness which harms the Vitamin D absorption, such as Celiac, chronic Pancreatitis, Cystic Fibrosis and IBS.
* people who have a chronic illness which harms Vitamin D metabolism, such as chronic hepatitis, kidney insufficiency and Nephrotic Syndrome.
* pregnant women.
* people who require prescribed medicine like steroids, anti-convulsion, and HIV treatments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People employed in three types of natural sunlight exposure.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-11